CLINICAL TRIAL: NCT07047794
Title: Relationship Between Scapula Position and Upper Extremity Joint Range of Motion, Strength and Performance in Children With Thoracic Hyperkyphosis
Brief Title: Scapula Position and Range of Motion, Strength and Performance in Thoracic Hyperkyphosis
Status: Completed | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Kubra Koce, Asst. Prof., Istinye University
Other Study IDs: 23/75
Record Dates: First submitted 2025-06-23; First posted 2025-07-02 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Hyperkyphosis
Keywords: thoracic hyperkyphosis; scapula; kinetic chain; upper extremity performance
MeSH Terms: conditions — Kyphosis | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — Children with thoracic hyperkyphosis between the ages of 7 and 14 who meet the inclusion criteria will be included in this study, which was conducted to examine the scapular position and its relationships with upper extremity joint range of motion, strength and performance in children with thoracic hyperkyphosis.

SUMMARY:
In the sagittal plane, the average kyphosis angle between the superior endplate of the T1 vertebra and the inferior endplate of the T12 vertebra is approximately 40 degrees. A thoracic spine angle greater than 45 degrees is defined as hyperkyphosis. The most common types of hyperkyphosis observed in juveniles and adolescents are Scheuermann's kyphosis, postural hyperkyphosis, and congenital hyperkyphosis.

Postural hyperkyphosis is the most prevalent form among these types. It results from the weakness of the muscles responsible for maintaining an upright posture and occurs due to external forces acting on the spine. The curvature of the spine in this condition is not rigid and can generally be corrected when the individual is asked to stand upright. Postural hyperkyphosis is typically seen during adolescence.

An increased thoracic kyphosis angle in postural hyperkyphosis can affect scapular kinematics, potentially leading to shoulder pathologies later in life, such as impingement syndrome, rotator cuff tendinopathy, rotator cuff tears, glenohumeral instability, and adhesive capsulitis. Additionally, hyperkyphosis can negatively affect body image and overall quality of life. If it begins in childhood and remains untreated, hyperkyphosis may persist into adulthood and contribute to increased healthcare expenditures. Given the growing prevalence of technology dependence and its association with rising hyperkyphosis incidence, early management of this deformity during juvenile and adolescent periods is essential in terms of both health and economic outcomes. In managing postural hyperkyphosis, it is important to address not only the angular correction of the deformity but also to consider the entire spine within the kinetic chain model.

The kinetic chain model is a biomechanical concept that defines the body as a system of interconnected segments. Any dysfunction within one segment of the kinetic chain can affect the quality of movement in both the upper and lower segments. The scapula serves as a foundation within this model, acting as a force transmitter that converts potential energy generated by muscles into kinetic energy in the upper extremity. Hyperkyphosis can lead to scapular protraction and downward rotation, disrupting the normal positioning of the scapula. As a result, joint range of motion, strength, and performance in the upper extremity may be negatively affected.

Studies in the literature have shown that scapular positioning and movements play a critical role in upper extremity function. However, no study has been found that specifically investigates the impact of altered scapular position on upper extremity performance in children with thoracic hyperkyphosis. Considering the increasing prevalence of thoracic hyperkyphosis in children due to rising technology addiction, and the potential for this deformity to contribute to upper extremity pathologies in adulthood, identifying its effects is crucial for improving children's physical performance and reducing future healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Being between 7-14 years old
* Thoracic kyphosis angle (Cobb) on lateral radiograph: ≥45˚ or kyphosis index ≤13

Exclusion Criteria:

* Those who have had major surgery or trauma related to the musculoskeletal system, especially the spine and upper extremities
* Difficulty in perceiving commands
* Rigid deformity in the spine (Scheuermann kyphosis)
* Congenital deformity

Ages: 7 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: Children with thoracic hyperkyphosis will be included in our study.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2025-06-23 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Sociodemographic Status | 4 weeks
  The sociodemographic status of the participants will be recorded with an evaluation form prepared by the researchers. Information on age, gender, dominant side, exercise habits will be questioned. Participants' privacy will be respected throughout the study, and no photographs will be taken.
Upper Extremity Range of Motion | 4 weeks
  Bilateral shoulder flexion, extension, abduction, elbow flexion, extension and wrist flexion and extension range of motion will be measured with a digital goniometer whose validity and reliability have been demonstrated.
Upper Extremity Muscle Strength | 4 weeks
  Bilateral trapezius upper-middle-lower fibers, serratus anterior, shoulder flexion, extension, abduction, elbow flexion, extension and wrist flexion and extension muscle strength will be measured with a myometer whose validity and reliability have been demonstrated.
Flexicurve Ruler | 4 weeks
  Flexicurve Ruler is a method that is preferred more than other methods because it is cheap, easy to use and has high validity and reliability. In our study, kyphosis curvatures will be measured with Flexicurve Ruler and kyphosis index will be calculated. Kyphosis index is the value found by dividing the width of the thoracic curvature by its length.
Wall-Occiput Distance | 4 weeks
  The increase in the thoracic kyphosis angle will be evaluated and recorded with the wall-occiput distance measurement. The distance between the occiput and the wall will be measured with a ruler while the individual to be tested stands in contact with the wall
Scapula Position | 4 weeks
  The Lateral Scapular Shift Test will be used to determine the scapula position in the 0, 45 and 90° abduction positions of the shoulder joint. Measurements of the scapular position will be made bilaterally in three test positions, between the spinous processes of the thoracic vertebrae in line with the inferior angle of the scapula.
Closed Kinetic Chain Upper Extremity Stability Test | 4 weeks
  Upper extremity will be used for strength, endurance and closed kinetic chain assessment. The test will be applied in a push-up position with the distance between the two hands set at 90 cm, then the number of repetitions completed within 15 seconds by extending one hand towards the other hand will be recorded.
Upper Extremity Y-Balance Test | 4 weeks
  It will be used to evaluate the balance, functionality and stability of the upper extremity and trunk. The evaluation will begin in a push-up position with both arms shoulder-width apart. Starting with the non-dominant hand, the maximum reachable distance in the medial, inferolateral and superolateral directions will be recorded
Medicine Ball Throwing Test | 4 weeks
  Upper extremity will be used to evaluate explosive power. In this test, the distance covered by throwing a 3 kg ball will be recorded
Height | 4 weeks
  The vertical distance from the top of the head to the heels of the individual. It will be measured in centimeters.
Weight | 4 weeks
  The mass of the individual's body in relation to gravity. It will be expressed in kilograms.
Waist Circumference | 4 weeks
  A circumferential measurement taken with a tape measure at the narrowest point of the waist, or at the midpoint between the lower margin of the last palpable rib and the top of the iliac crest, to assess abdominal fat distribution. It will be measured in centimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided